CLINICAL TRIAL: NCT04735393
Title: A Multi-Center, Double-Masked, Randomized, Vehicle-Controlled, Parallel-Group Clinical Trial Evaluating the Safety of 0.25% Reproxalap Ophthalmic Solution in Subjects With Dry Eye Disease
Brief Title: A Multi-Center, Double-Masked, Randomized, Vehicle-Controlled, Parallel-Group Clinical Trial Evaluating the Safety of Reproxalap Ophthalmic Solution in Subjects With Dry Eye Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aldeyra Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ADX-102-DED-021
Record Dates: First submitted 2021-01-25; First posted 2021-02-03 (Actual); Results first posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-01

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Reproxalap (0.25%) for six weeks (Experimental): Reproxalap four times daily (QID) for four weeks followed by two times daily (BID) for two weeks
  Interventions: Drug: Reproxalap Ophthalmic Solution (0.25%)
- Vehicle for six weeks (Placebo Comparator): Vehicle QID for four weeks followed by BID for two weeks
  Interventions: Drug: Placebo Comparator
- Reproxalap (0.25%) for 12 months (Experimental): Reproxalap (0.25%) QID for four weeks followed by BID for 11 months
  Interventions: Drug: Reproxalap Ophthalmic Solution (0.25%)
- Vehicle for 12 months (Placebo Comparator): Vehicle QID for four weeks followed by BID for 11 months
  Interventions: Drug: Placebo Comparator

INTERVENTIONS:
Drug: Reproxalap Ophthalmic Solution (0.25%) — Reproxalap Ophthalmic Solution (0.25%) administered for six weeks (QID for four weeks then BID for two weeks).
  Arms: Reproxalap (0.25%) for six weeks
Drug: Placebo Comparator — Vehicle Ophthalmic Solution administered for six weeks (QID for four weeks then BID for two weeks).
  Arms: Vehicle for six weeks
Drug: Reproxalap Ophthalmic Solution (0.25%) — Reproxalap Ophthalmic Solution (0.25%) administered for one year (QID for four weeks then BID for 11 months).
  Arms: Reproxalap (0.25%) for 12 months
Drug: Placebo Comparator — Vehicle Ophthalmic Solution administered for one year (QID for four weeks then BID for 11 months).
  Arms: Vehicle for 12 months

SUMMARY:
A Multi-Center, Double-Masked, Randomized, Vehicle-Controlled, Parallel-Group Clinical Trial Evaluating the Safety of 0.25% Reproxalap Ophthalmic Solution in Subjects with Dry Eye Disease

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age (either gender and any race);
* Reported history of dry eye for at least 6 months prior to Visit 1;
* History of use or desire to use eye drops for dry eye symptoms within 6 months of Visit 1.

Exclusion Criteria:

* Clinically significant slit lamp findings at Visit 1 that may include active blepharitis, meibomian gland dysfunction (MGD), lid margin inflammation, or active ocular allergies that require therapeutic treatment, and/or in the opinion of the investigator may interfere with study parameters;
* Diagnosis of an ongoing ocular infection (bacterial, viral, or fungal), or active ocular inflammation at Visit 1;
* Contact lens use within 7 days of Visit 1 or anticipate using contact lenses during the trial;
* Eye drop use within 2 hours of Visit 1;
* Previous laser-assisted in situ keratomileusis (LASIK) surgery within the last 12 months;
* Cyclosporine 0.05% or 0.09% or lifitegrast 5.0% ophthalmic solution within 90 days of Visit 1;
* Planned ocular and/or lid surgeries over the study period or any ocular surgery within 6 months of Visit 1;
* Temporary punctal plugs during the study that have not been stable within 30 days of Visit 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 757 (Actual)
Dates: Start 2021-01-26 (Actual); Primary Completion 2022-10-11 (Actual); Study Completion 2022-10-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Andover Eye Associates, Andover, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The 6-week safety population are subjects randomized and treated in either the 6-week or 12-month cohort. The 12-month safety population are subjects randomized and treated in the 12-month cohort. There was a total of 757 randomized subjects in the trial. There were 6 subjects randomized and not dosed.
Groups:
- Reproxalap: Reproxalap was administered four times daily for four weeks followed by two times daily for either two weeks or 11 months.
- Vehicle: Vehicle was administered four times daily for four weeks followed by two times daily for either two weeks or 11 months.
Period: Overall Study
Arm/Group | Reproxalap | Vehicle
Started | 504 | 253
As Treated | 501 (There were 504 subjects assigned to reproxalap. Three subjects were assigned to reproxalap and never dosed. One subject was assigned to reproxalap and were also dosed with vehicle.) | 250 (There were 253 subjects assigned to vehicle. Three subjects were assigned to vehicle and never dosed. Two subjects were assigned to vehicle and were also dosed with reproxalap.)
Completed | 273 | 161
Not Completed | 231 | 92
Not completed — Lost to Follow-up | 46 | 24
Not completed — Physician Decision | 2 | 1
Not completed — Not Detailed | 1 | 2
Not completed — Withdrawal by Subject | 71 | 28
Not completed — Adverse Event | 56 | 7
Not completed — Protocol Violation | 6 | 1
Not completed — Trial terminated by Sponsor | 49 | 29

BASELINE CHARACTERISTICS:
Population: 6-week safety population
Groups:
- Reproxalap (6-week): Reproxalap was administered four times daily for four weeks followed by two times daily for two weeks.
- Vehicle (6-week): Vehicle was administered four times daily for four weeks followed by two times daily for two weeks.
- Total: Total of all reporting groups
Arm/Group | Reproxalap (6-week) | Vehicle (6-week) | Total
Number analyzed (Participants) | 503 | 251 | 754
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 336 | 165 | 501
  >=65 years | 167 | 86 | 253
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.7 (15.8) | 56.9 (15.8) | 56.0 (15.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 356 | 176 | 532
  Male | 147 | 75 | 222
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 154 | 75 | 229
  Not Hispanic or Latino | 349 | 176 | 525
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 28 | 15 | 43
  Asian | 68 | 42 | 110
  Black or African American | 54 | 26 | 80
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  White | 343 | 162 | 505
  Other | 1 | 2 | 3
  Multiple | 8 | 4 | 12

OUTCOME MEASURES:

1. Primary Outcome: Treatment-Emergent Serious Adverse Events (TE-SAEs) of Visual Acuity Decrease
Description: The proportion of 6-week safety population subjects that experience at least one visual acuity TE-SAE decrease (defined as an increase of 0.22 or greater in logMAR score) categorized as probably or definitely related to test article.
Time Frame: Safety assessment period (six weeks)
Population: 6-week safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Reproxalap | Vehicle
Number analyzed (Participants) | 503 | 251
Participants | 0 | 0

2. Primary Outcome: TE-SAEs of Increase in Intraocular Pressure
Description: The proportion of 6-week safety population subjects that experience at least one intraocular pressure TE-SAE (increase from baseline of greater than or equal to 10 mmHg and intraocular pressure of greater than 25 mmHg) categorized as probably or definitely related to test article.
Time Frame: Safety assessment period (six weeks)
Population: 6-week safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Reproxalap | Vehicle
Number analyzed (Participants) | 503 | 251
Participants | 0 | 0

3. Primary Outcome: TE-SAEs of the Cornea
Description: The proportion of 6-week safety population subjects that experience at least one cornea-related TE-SAE (detected via slit-lamp examination) categorized as probably or definitely related to test article.
Time Frame: Safety assessment period (six weeks)
Population: 6-week safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Reproxalap | Vehicle
Number analyzed (Participants) | 503 | 251
Participants | 0 | 0

4. Primary Outcome: TE-SAEs of the Retina
Description: The proportion 6-week safety population subjects that experience at least one retinal TE-SAE (detected via fundoscopy) categorized as probably or definitely related to test article.
Time Frame: Safety assessment period (six weeks)
Population: 6-week safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Reproxalap | Vehicle
Number analyzed (Participants) | 503 | 251
Participants | 0 | 0

5. Post Hoc Outcome: Change From Baseline in Visual Acuity
Description: Overall change from baseline in visual acuity logMAR score. Visual acuity values were averaged across both eyes for each participant.
Time Frame: Efficacy assessment period (12 months)
Population: 12-month primary safety analysis population
Measure: Least Squares Mean (Standard Error); unit: LogMAR
Units Other Than Participants: eyes
Groups:
- Reproxalap: Reproxalap was administered four times daily for four weeks followed by two times daily for 11 months.
- Vehicle: Vehicle was administered four times daily for four weeks followed by two times daily for 11 months.
Arm/Group | Reproxalap | Vehicle
Number analyzed (Participants) | 296 | 145
Number analyzed (eyes) | 592 | 290
LogMAR | -0.030 (0.0035) | -0.016 (0.0046)

6. Primary Outcome: TE-SAEs of Visual Acuity Decrease
Description: The proportion of 12-month safety population subjects that experience at least one visual acuity TE-SAE (defined as an increase of 0.22 or greater in logMAR score) categorized as probably or definitely related to test article.
Time Frame: Safety assessment period (12 months)
Population: 12-month safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Reproxalap | Vehicle
Number analyzed (Participants) | 299 | 148
Participants | 0 | 0

7. Primary Outcome: TE-SAEs of Increase in Intraocular Pressure
Description: The proportion of 12-month safety population subjects that experience at least one intraocular pressure TE-SAE (increase from baseline of greater than or equal to 10 mmHg and intraocular pressure of greater than 25 mmHg) categorized as probably or definitely related to test article.
Time Frame: Safety assessment period (12 months)
Population: 12-month safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Reproxalap | Vehicle
Number analyzed (Participants) | 299 | 148
Participants | 0 | 0

8. Primary Outcome: TE-SAEs of the Cornea
Description: The proportion of 12-month safety population subjects that experience at least one cornea-related TE-SAE (detected via slit-lamp examination) categorized as probably or definitely related to test article.
Time Frame: Safety assessment period (12 months)
Population: 12-month safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Reproxalap | Vehicle
Number analyzed (Participants) | 299 | 148
Participants | 0 | 0

9. Primary Outcome: TE-SAEs of the Retina
Description: The proportion 12-month safety population subjects that experience at least one retinal TE-SAE(detected via fundoscopy) categorized as probably or definitely related to test article.
Time Frame: Safety assessment period (12-months)
Population: 12-month safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Reproxalap | Vehicle
Number analyzed (Participants) | 299 | 148
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Safety assessment period (6 weeks or 12 months)
Groups:
- Reproxalap (12-month): Reproxalap was administered four times daily for four weeks followed by two times daily for 11 months.
- Vehicle (12-month): Vehicle was administered four times daily for four weeks followed by two times daily for 11 months.
Arm/Group | Reproxalap (6-week) | Vehicle (6-week) | Reproxalap (12-month) | Vehicle (12-month)
All-Cause Mortality (participants affected / at risk) | 0/503 | 0/251 | 0/299 | 2/148
Serious Adverse Events (participants affected / at risk) | 0/503 | 0/251 | 3/299 | 5/148
Other Adverse Events (participants affected / at risk) | 205/503 | 8/251 | 127/299 | 3/148
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reproxalap (6-week) (N=503) | Vehicle (6-week) (N=251) | Reproxalap (12-month) (N=299) | Vehicle (12-month) (N=148)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — The SAE was deemed not related to study drug.
COVID-19 Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — The SAE was deemed not related to study drug.
Unknown cause of death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — The SAE was deemed not related to study drug.
Premature ventricular contractions (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — The SAE was deemed not related to study drug.
Unstable Angina (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — The SAE was deemed not related to study drug.
Worsening coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Right tonsil squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — The SAE was deemed not related to study drug.
Worsening of chronic back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — The SAE was deemed not related to study drug.
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — The SAE was deemed not related to study drug.
Supraventricular Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — The SAE was deemed not related to study drug.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reproxalap (6-week) (N=503) | Vehicle (6-week) (N=251) | Reproxalap (12-month) (N=299) | Vehicle (12-month) (N=148)
General disorders and administration site conditions (General disorders) | 205 (205) | 8 (8) | 127 (127) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-16): https://cdn.clinicaltrials.gov/large-docs/93/NCT04735393/Prot_SAP_000.pdf